CLINICAL TRIAL: NCT03297736
Title: Improved Otologic Implants on Demand Intraoperatively With 3D CAD/CAM Autografts
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nitinetics LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Device Feasibility
Other Study IDs: 3D CAD/CAM
Record Dates: First submitted 2017-09-13; First posted 2017-09-29 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Middle Ear Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Subjects receive the control device.
  Interventions: Device: Control device
- Investigational device (Experimental): Subject receives the 3D CAD/CAM autograft prosthesis implant.
  Interventions: Device: 3D CAD/CAM autograft prosthesis

INTERVENTIONS:
Device: 3D CAD/CAM autograft prosthesis — Surgical ossicular reconstruction with the experimental autograft prosthesis created using 3D subtraction CAD/CAM.
  Arms: Investigational device
Device: Control device — Surgical ossicular reconstruction with the standard available middle ear prosthesis.
  Arms: Control

SUMMARY:
Prospectively analyze the use of 3D subtraction CAD/CAM in the operating room environment. Study participants, requiring middle ear surgery and ossicular reconstruction, will be implanted with one of two middle ear implants. The rationale is to complete a pilot study of the technology with a small number of designs. Each implant will be commonly used, in the public domain, and recreated by the CAD/CAM software.

DETAILED DESCRIPTION:
Conventional middle ear prosthetic prosthetics, including total ossicular replacement prostheses (TORPs) and partial ossicular replacement prostheses (PORPs) are expensive, require large inventories for otologic surgery services, and carry the risk of extrusion or rejection. Autologous bone and cartilage can be used for many of these applications, but it requires expensive operating room time for carving to the appropriate shape and size.

The above considerations led to the concept of subtractive 3D CAD/CAM (computer assisted design/computer assisted manufacture) to produce accurate bone and cartilage autografts on demand in the operating room. Such a technology is hypothesized to save money by reducing operating room time, and reducing the need for expensive inventories of various shapes, sizes, and types of prosthetic devices. Since autologous materials are hypothesized to be less likely to extrude or cause other problems such as infection, this could also reduce costs.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age with middle ear disease requiring surgical ossicular reconstruction

Exclusion Criteria:

* congenital anomalies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-03-01 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Cost savings | perioperative
  operative costs compared between treatment groups utilizing total operative time in minutes

SECONDARY OUTCOMES:
Number of participants with treatment related adverse events as assessed by CTCAE v4.0 | 6 months
  infectious process involving the use of a medical device
ABG | preoperative; 6weeks, 3 months, and 6 months postoperatively.
  mean air-bone gap assessed and compared between treatment groups for statistical significance
Number of participants that experience device rejection | 6 months
  rejection of device/prosthesis

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Knox, M.D., J.D., Principal Investigator — Nitinetics LLC
Locations (1):
- University of Florida-Jacksonville, Jacksonville, Florida, United States